CLINICAL TRIAL: NCT01465217
Title: Text Messaging to Improve Hypertension Medication Adherence in African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lorraine Buis, Assistant Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R21HS019092-01 (AHRQ)
Record Dates: First submitted 2011-11-01; First posted 2011-11-04 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Hypertension
Keywords: medication adherence; African Americans
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- text message medication reminders (Experimental)
  Interventions: Behavioral: text message medication reminders
- control (No Intervention)

INTERVENTIONS:
Behavioral: text message medication reminders — daily medication reminders for one month
  Arms: text message medication reminders

SUMMARY:
Uncontrolled high blood pressure (HBP) is a major public health concern and leading cause of cardiovascular disease worldwide. The HBP crisis is particularly onerous to African Americans as they are disproportionately more susceptible to HBP than non-Hispanic White Americans. Poor adherence to prescribed medication regimens is a major problem, as only about half of patients who have been diagnosed with hypertension adhere to prescribed medications. Mobile phones and text messages are becoming widely integrated into routine daily life and may offer a simple and non-labor intensive strategy for improving the quality of medication management through enhancing medication adherence. This proposed research will be conducted in two distinct phases addressing three specific aims. For Specific Aim 1 (Phase I), the investigators propose to conduct focus groups with participants from the investigators target population in order to obtain feedback to guide the development of a mobile phone text message system that seeks to improve adherence to antihypertensive medications. For Specific Aim 2 (Phase II), the investigators propose to pilot test the newly developed text message intervention with a randomized controlled trial. For Specific Aim 3 (Phase II), the investigators propose to ascertain participant perceptions of intervention effectiveness and satisfaction in order to guide further system refinement. In Phase I, African Americans with uncontrolled hypertension (n=24-32) will be recruited to take part in one of four focus groups that will help guide the development of the text message intervention. In Phase II, African Americans with uncontrolled hypertension will be randomized to receive usual care (n=30) vs. the text message intervention (n=30). The primary outcome in this pilot will be change in medication adherence at one month follow-up; secondary outcomes include change in medication self-efficacy and systolic and diastolic blood pressure at one month follow-up, as well as participant satisfaction with the text message intervention. The proposed research will utilize the Wayne State University (WSU) Center for Urban Studies to conduct high quality and professionally run focus groups, the WSU Division of Computing and Information Technology's Broadcast Message Service infrastructure for the delivery of text messages, the WSU Center for Health Research for statistical analysis and grant management assistance, and a diverse study team from a variety of disciplinary backgrounds at WSU. As a result, the proposed research leverages the considerable local resources to investigate an innovative and much needed intervention for this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as African American/Black
* be >18 years
* have a diagnosis of HBP based on ICD-9 codes
* have uncontrolled hypertension on two successive clinic visits prior to screening (clinic SBP > 140 mm Hg, DBP > 90 mm Hg or SBP > 130, DBP > 80 for those with diabetes or kidney disease) as documented in the medical record
* be taking at least one antihypertensive medication
* own a cell phone capable of receiving and sending text messages
* be able to pay for and obtain hypertension medication
* English speaking
* willing to attend two data collection visits in Detroit, MI

Exclusion Criteria:

* receiving hemodialysis
* admits to planning to terminate cell phone contract during the next one month
* compliance risk (i.e., self-reported illicit drug use and/or alcohol abuse as measured by a score of >2 for CAGE questions
* health literacy less than third grade reading level
* other major health problems (e.g., terminal stage of cancer, advanced liver disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-03; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
medication adherence | one month

SECONDARY OUTCOMES:
medication self efficacy | one month
blood pressure | one month

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine R Buis, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Derived] Buis L, Hirzel L, Dawood RM, Dawood KL, Nichols LP, Artinian NT, Schwiebert L, Yarandi HN, Roberson DN, Plegue MA, Mango LC, Levy PD. Text Messaging to Improve Hypertension Medication Adherence in African Americans From Primary Care and Emergency Department Settings: Results From Two Randomized Feasibility Studies. JMIR Mhealth Uhealth. 2017 Feb 1;5(2):e9. doi: 10.2196/mhealth.6630. PMID 28148474
- [Derived] Buis LR, Artinian NT, Schwiebert L, Yarandi H, Levy PD. Text Messaging to Improve Hypertension Medication Adherence in African Americans: BPMED Intervention Development and Study Protocol. JMIR Res Protoc. 2015 Jan 2;4(1):e1. doi: 10.2196/resprot.4040. PMID 25565680